CLINICAL TRIAL: NCT03490084
Title: Impacts on Health Outcomes and Resources Utilization of Hospital-at-home for Elderly Patients With Multiple Myeloma
Acronym: PAMM-HAD1
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: K160917J; 2017-A03219-44 (Registry Identifier: IDRCB)
Record Dates: First submitted 2018-02-26; First posted 2018-04-06 (Actual); Last update posted 2023-08-28 (Actual); Status verified 2023-08

CONDITIONS: Multiple Myeloma
Keywords: multiple myeloma; elderly patients; health outcomes; hospital-at-home; day hospitalization; quality of life; medico-economic evaluation; qualitative study
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Association of day hospitalization with hospital-at-home: Patients receive the first administration of chemotherapy through day hospitalization in the hematology department, then 3 weekly administrations of chemotherapy at home.
  Interventions: Other: Association of day hospitalization with hospital-at-home
- Day hospitalization exclusively: Patients receive 4 weekly administrations of chemotherapy through day hospitalization in the hematology department.
  Interventions: Other: Day hospitalization exclusively

INTERVENTIONS:
Other: Association of day hospitalization with hospital-at-home — Patients receive the first administration of chemotherapy through day hospitalization in the hematology department, then 3 weekly administrations of chemotherapy at home.
  Groups: Association of day hospitalization with hospital-at-home
Other: Day hospitalization exclusively — Patients receive 4 weekly administrations of chemotherapy through day hospitalization in the hematology department.
  Groups: Day hospitalization exclusively

SUMMARY:
The study aims to compare the overall survival adjusted to quality of life of 2 groups of patients with multiple myeloma, depending on the type of care: (1) day hospitalization exclusively or (2) day hospitalization combined with hospital-at-home.

As secondary objectives, the study aims to compare the impacts of the two types of care organization on:

* the survival of patients and response to treatments according to criteria of the International Myeloma Working Group,
* psychological status of patients,
* specific toxicity related to treatment used (haematological and infectious toxicity, neurotoxicity, ...),
* health outcomes,
* the caregiver's burden,

This study is combined with a qualitative study about the incentives and the barriers, and in order to set up the patient's typology.

DETAILED DESCRIPTION:
Multiple myeloma, a malignant blood disease with about 5000 new cases diagnosed annually in France, essentially in the elderly population, is associated with alteration of quality of life resulting from pathology and therapies.

Multiples cycles of chemotherapies are administered in a regular manner, as outpatient treatment or day hospitalization.

In this study aiming to explore the impacts on health outcomes and resources utilization of hospital-at-home for elderly patients with multiple myeloma, all patients will be treated by 4 standardized protocols of treatment including bortezomib by subcutaneous administration.

9 centers will participate to the study. The study will not change the usual practices of care of these centers:

* 6 centers organize patient care through day hospitalization combined with hospital-at-home,
* 3 other centers rely exclusively on day hospitalization.

The study will target overall the inclusion of 300 patients for the 9 centers and 70 participants (35 for each arm: 10 patients, 10 caregivers, 15 from healthcare team) for the qualitative study.

The individual follow up of each patient will last 12 months. The patient's vital status will be documented at the 24th month.

ELIGIBILITY:
Inclusion Criteria:

* Patient > 65 years;
* Resident of the departments in Île-de-France region (75, 92, 93 and 94);
* Symptomatic multiple myeloma (relapsed or no);
* Patient planned to receive one of the following chemotherapy protocols including bortezomib (VELCADE®): VMP (Velcade, Melphalan, Prednisone), VCD (Velcade, Cyclophosphamide, Dexamethasone), VelDex (Velcade, Dexamethasone), VRD (Velcade, Revlimid, Dexamethasone);
* Ineligible for autologous hematopoietic stem-cell transplantation (ASCT);
* Covered by a health insurance;
* Patient who does not oppose to the use of his/her medical data for the purpose of clinical research.
* Adult patients under guardianship will can be enrolled in the study, a consent of tutor is needed completed by patient's consent.

Exclusion Criteria:

* Resident of the departments of 77, 78 and 91 in Île-de-France region;
* Asymptomatic myeloma;
* Life expectancy < 6 months;
* Patient does not understand French language.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patient aged > 65 years, with symptomatic multiple myeloma, ineligible for autologous hematopoietic stem-cell transplantation, planned to undergo treatments including bortezomib.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-02-25 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Change in Quality of life using questionnaires EORTC QLQ-30 | At baseline, at the 6th month and the 12th month
  Comparison of quality of life using questionnaires EORTC QLQ-30.
Change in Quality of life using questionnaires EORTC QLQ-MY20 | At baseline, at the 6th month and the 12th month
  Comparison of quality of life using questionnaires EORTC QLQ-MY20.

SECONDARY OUTCOMES:
Survival | At the 1st day of each chemotherapy cycle (each cycle varying between 28 and 35 days)
  All patients will be evaluated in order to collect the following data:
  * death and causality with multiple myeloma, treatments;
  * progression or relapse according to criteria of International Myeloma Working Group;
  * survival without progression, full or partial remission.
Multidimensional evaluation of home care | At baseline, at the 6th month
  RAI-HC (Resident Assessment Instrument Home Care) will be used at home. Multidimensional evaluation involves 19 areas such as sociodemographic, environmental and clinical endpoints with psychological status, cognitive status, morbidity and medication compliance defined by validated synthetic clinical scales.
Toxicity of treatment | At baseline, at each evaluation of response to therapy, at the 6th month and the 12th month
  This evaluation will be performed for all patients with the National Cancer Institute Common Terminology Criteria for Adverse Events (CRCAE version 3.0).
family quality of life | At baseline, at the 6th month and the 12th month
  Family quality of life will be evaluated with Zarit Burden Inventory
Total Cost | At the end of study: 3 years
  The following costs will be collected: hospitalization, home care, transport, biological exams, costs of chemotherapy (bortezomib) as well as indirect costs such as paid sick leave and salary of caregiver at home.
Fate-to-face interview with patients, caregivers and healthcare staff | At baseline, at the 6th month and the 12th month
  The assessment criteria are the quality care, the continuity of care, the coordination between the care actors, the information transmission, the incentives and the barriers according to the forms of hospitalization.

CONTACTS AND LOCATIONS:
Overall Officials: Bénédicte MITTAINE-MARZAC, PharmD, Study Chair — Hospitalisation à domicile (HAD), APHP; Matthieu de STAMPA, MD, Study Director — Hospitalisation à domicile (HAD), APHP
Locations (1):
- HAD, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No